CLINICAL TRIAL: NCT05462704
Title: Double-blind Placebo-controlled Multicenter Randomized Trial of Intravenous Versus Oral Iron for Treating Iron-Deficiency Anemia in Pregnancy
Brief Title: Intravenous Versus Oral Iron for Treating Iron-Deficiency Anemia in Pregnancy
Acronym: IVIDA2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: Hasbro Children's Hospital (Other); University of Michigan (Other); Washington University School of Medicine (Other); University of Utah (Other); University of Alabama at Birmingham (Other); Oregon Health and Science University (Other); GNP Research at Heme-on-Call (Unknown)
Responsible Party: Principal Investigator, Methodius Tuuli, Professor and Chair of Obstetrics and Gynecology, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00060930
Record Dates: First submitted 2022-05-15; First posted 2022-07-18 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Iron Deficiency Anemia; Pregnancy
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric derisomaltose; ferrous sulfate; Iron-Dextran Complex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will receive matching ferrous sulfate or placebo formulate to appear and taste similar. They will also each receive an infusion of 1000mg ferric derisomaltose in 250ml of normal saline or 250ml of normal saline only, camouflaged in an opaque intravenous bag and tubing covers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- IV Iron (Experimental): Participants assigned to the IV iron group will receive a single IV infusion of 1000 mg ferric derisomaltose (Monoferric, Pharmacosmos Therapeutics Inc., Morristown, NJ) in 250 mL given over 20 minutes and daily placebo tablets until delivery.
  Interventions: Drug: Ferric derisomaltose
- Oral Iron (Active Comparator): Participants assigned to the oral iron group will receive a single 250 mL IV normal saline infusion given over 20 minutes and 325mg tablets of ferrous sulfate (65 mg of elemental iron) to be taken until delivery.
  Interventions: Drug: Ferrous sulfate

INTERVENTIONS:
Drug: Ferric derisomaltose — Participants assigned to the IV iron group will receive a single IV infusion of 1000 mg ferric derisomaltose (Monoferric, Pharmacosmos Therapeutics Inc., Morristown, NJ) in 250 mL given over 20 minutes.
  Other Names: Monoferric
  Arms: IV Iron
Drug: Ferrous sulfate — 325mg ferrous sulfate tablets (65 mg of elemental iron), 1 to 3 orally per day.
  Other Names: Ferosul
  Arms: Oral Iron

SUMMARY:
Double blind, placebo controlled, multicenter randomized trial in pregnant women in the U.S. (N=300) to test the central hypothesis that IV iron in pregnant women with IDA (Hb<11 g/dL and ferritin<30 ng/mL) at 13 - 30 weeks will be effective, safe and cost-effective in reducing severe maternal morbidity-as measured by maternal anemia at delivery-and will also improve offspring neurodevelopment.

DETAILED DESCRIPTION:
Iron-deficiency anemia (IDA) is a common, undertreated problem in pregnancy. According to data from the U.S. National Health and Nutrition Examination Survey (NHANES), 25% of pregnant women in the U.S. have iron deficiency, with rates of 7%, 24%, and 39% in the first, second, and third trimesters, respectively. The prevalence of IDA is estimated at 16.2% overall and up to 30% at delivery. Iron deficiency is associated with significant adverse maternal and fetal outcomes including blood transfusion, cesarean delivery, depression, preterm birth, and low birth weight. Moreover, iron-deficient mothers are at risk of delivering iron-deficient neonates who, despite iron repletion, remain at risk for delayed growth and development. While treatment with iron supplementation is recommended during pregnancy, questions remain about the optimal route of delivery. Oral iron therapy, the current standard, is often suboptimal: up to 70% of patients experience significant gastrointestinal side effects (nausea, constipation, diarrhea, indigestion, and metallic taste) that prevent adherence to treatment, resulting in persistent anemia. Intravenous (IV) iron is an attractive alternative because it mitigates the adherence and absorption challenges of oral iron. However, IV iron costs more, and there are historical concerns about adverse reactions.

The American College of Obstetricians and Gynecologists (ACOG) recommends oral iron for the treatment of IDA in pregnancy, with IV iron reserved for the restricted group of patients. Our preliminary data show that this approach leads to 30% of patients with persistent IDA at delivery and an associated 3 to 6-fold increased risk of peripartum blood transfusion. ACOG's preferential recommendation of oral iron is based on paucity of data on the benefits and safety of IV iron, compared with oral iron, in pregnancy. Our published systematic review and meta-analysis showed that IV iron is associated with greater increase in maternal hemoglobin (Hb), but most of the primary trials were conducted in developing countries, included small sample sizes (50 - 252), and did not assess meaningful maternal and neonatal outcomes. The current Cochrane review noted that despite the high incidence and disease burden associated with IDA in pregnancy, there is paucity of quality trials assessing clinical maternal and neonatal effects of iron administration in women with anemia. The authors called for "large, good quality trials assessing clinical outcomes." The only large randomized trial of IV versus oral iron, conducted in India, showed no difference in a maternal composite outcome, but it is limited by use of iron sucrose which required five infusions, resulting in a wide range of iron doses (200 - 1600 mg). In addition, the primary composite outcome included some components not directly related to anemia. In contrast, our pilot trial of a single infusion of 1000 mg of IV low molecular weight iron dextran in pregnant women in the U.S. with moderate-to-severe IDA significantly reduced the rate of maternal anemia at delivery and showed promise for improving maternal morbidity by reducing rates of blood transfusion.

This is the first definitive double blind, placebo controlled, multicenter randomized trial in pregnant women in the U.S. (N=300) to test the central hypothesis that IV iron in pregnant women with IDA (Hb<11 g/dL and ferritin<30 ng/mL) at 13 - 30 weeks will be effective, safe and cost-effective in reducing severe maternal morbidity-as measured by maternal anemia at delivery-and will also improve offspring neurodevelopment. A multidisciplinary team of investigators in the U.S., will pursue the following specific aims:

Primary Aim: Evaluate the effectiveness and safety of IV iron, compared with oral iron, in reducing the rate of anemia at delivery in pregnant women with IDA.

Secondary Aim 1: Estimate the cost-effectiveness of IV iron , compared with oral iron, in pregnant women with IDA as measured by incremental cost per Quality Adjusted Life-year (QALY).

Secondary Aim 2: Assess the effect of IV iron, compared with oral iron, on offspring brain myelin content and neurodevelopment.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between the ages of 18-45
* Singleton gestation
* Iron-deficiency anemia (serum ferritin <30ng/mL and Hb<11 g/dL)
* At 13-30 weeks gestation
* Plan to deliver at participating hospital

Exclusion Criteria:

* Non-iron-deficiency anemia e.g thalassemia, sickle cell disease, B12 or folate deficiency, hypersplenism.
* Malabsorptive syndrome, inflammatory bowel disease, gastric bypass, or sensitivity to oral or IV iron
* Multiple gestation
* Inability or unwillingness to provide informed consent
* Inability to communicate with members of the study team, despite the presence of an interpreter
* Planned delivery at a non-study affiliated hospital

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients must be pregnant in order to participate
Enrollment: 300 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of maternal anemia (hgb<11mg/dL) at delivery | Within 24 hours of admission to inpatient obstetrics unit for delivery of infant
  Hemoglobin <11mg/dL on admission to inpatient obstetrics unit for labor and delivery

SECONDARY OUTCOMES:
Concentration of maternal hemoglobin at delivery | Within 24 hours of admission to inpatient obstetrics unit for delivery of infant
  Hemoglobin on admission to inpatient obstetrics unit for labor and delivery
Rate of maternal blood transfusion at delivery | Delivery to 7 days postpartum
  Maternal blood transfusion from delivery to 7 days postpartum
Concentration of maternal ferritin at delivery | Within 24 hours of admission to inpatient obstetrics unit for delivery of infant
  Maternal ferritin on admission to inpatient obstetrics unit for labor and delivery
Concentration of maternal hemoglobin postpartum day 1 | On day after participant delivered her infant; postpartum day 1
  Maternal hemoglobin on postpartum day 1
Rate of cesarean delivery | Once at infant delivery
  Cesarean delivery for any indication in patients without prior cesarean deliveries
Rate of severe infusion adverse events | 2 days after intravenous iron or placebo infusion
  Safety and tolerability
Rate of mild medication adverse events | 4 weeks after initiation of oral iron or placebo
  Safety and tolerability
Edinburgh Perinatal Depression Scale score | At randomization (baseline) and at 4-6 weeks postpartum
  Edinburgh Perinatal Depression Scale score. Minimum score 0, maximum score 30, higher scores indicate worse depressive symptoms.
Maternal EuroQol Group Quality-of-Life Questionnaire score | At 6 weeks postpartum by phone or in person
  Maternal EuroQol Group Quality-of-Life Questionnaire (EQ-5D-5L). Minimum score 11111 (full health), maximum score 55555 (worst health), higher scores indicate worse quality of life.
Rate of Maternal infection | From initiation of treatment until 6 weeks postpartum
  Any infection diagnosed from initiation of treatment until 6 weeks postpartum
Rate of Composite Maternal Complications | At 6 weeks postpartum
  Maternal mortality or any one of several maternal morbidities
Gestational age at delivery | At delivery
  Gestational age at delivery
Rate of preterm birth at less then 37 weeks | At delivery
  Preterm birth; gestational age at delivery at less than 37 weeks (spontaneous or indicated)
Rate of Neonatal Intensive Care Unit Admission | At birth through through 30 days from birth
  Admission to the neonatal intensive care unit for any indication
Neonatal birth weight | At birth
  Infant birth weight
Concentration of umbilical artery pH | At birth
  Concentration of umbilical artery pH from umbilical cord gases from infant umbilical cord segment at birth
Concentration of umbilical artery bicarbonate | At birth
  Concentration of umbilical artery bicarbonate from umbilical cord gases from infant umbilical cord segment at birth
Concentration of umbilical artery base excess | At birth
  Concentration of base excess from umbilical cord gases from infant umbilical cord segment at birth
Concentration of umbilical artery lactate | At birth
  Concentration of umbilical artery lactate from umbilical cord gases from infant umbilical cord segment at birth
Concentration of neonatal hemoglobin | At birth
  Concentration of neonatal hemoglobin from umbilical cord blood at birth or first neonatal complete blood count
Concentration of neonatal ferritin | At birth
  Concentration of neonatal ferritin from umbilical cord blood at birth or first neonatal blood draw
Neonatal Apgar scores | At 1 minute and 5 minutes of life
  Apgar scores at 1 and 5 minutes of life. Minimum score 0, maximum score 10, higher scores indicate better well being.
Rate of composite neonatal complication | Through 30 days from birth
  Neonatal mortality or any one of several neonatal morbidities
Concentration of child brain myelin | At an average of 6 months and 36 months
  Concentration of infant brain myelin from magnetic resonance imaging
Child Mullen Scale of Early Learning Score | At an average of 6 months and 36 months
  Mullen Scale of Early Learning Score as percentile. Minimum score 1, maximum score 99, higher scores indicate better neurodevelopment.

CONTACTS AND LOCATIONS:
Overall Officials: Methodius Tuuli, MD, MPH, MBA, Principal Investigator — Women and Infants Hospital of Rhode Island
Locations (8):
- United States (8):
  - University of Alabama Medical Center, Birmingham, Alabama
  - GNP Research at Heme-on-Call, Miami, Florida
  - Michigan University Medical Center, Ann Arbor, Michigan
  - Washington University Medical Center, St Louis, Missouri
  - Oregon Health and Sciences Uiversity Medical Center, Portland, Oregon
  - Hasbro Children's Hospital, Providence, Rhode Island
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Utah Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected from human subjects and will be shared according to NIH guidelines. The investigators are committed to the sharing of final data, being mindful that the rights and privacy of people who participate in research must be protected at all times. The investigators will make a complete study dataset available for sharing. The investigators will have a description of study dataset, including code books, meta-data related to the dataset, and documented programming code used for creating the final study population, for creating variables, and for conducting all outcomes analyses. The investigators will remain HIPAA compliant, and therefore any datasets resulting from participants will be free of any identifiers that would permit linkages to individual research participants and variables that could lead to deductive disclosure of individual subjects.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 5 years after completion of study
Access Criteria: The investigators will make the data and associated documentation available to users under a data-sharing agreement that provides for commitment to: a) using the data only for research purposes and not to identify any individual participant; b) securing the data using appropriate computer technology; and c) destroying or returning the data after analyses are completed. Timelines for distribution of data will vary depending on any required restrictions as mentioned above. Data may be distributed by a number of electronic methods, including web-based databases, datasets, and spreadsheets, or via electronic media such as compact discs.